CLINICAL TRIAL: NCT02581319
Title: Clinical Conditions and Prevalence of Periodontopathogens in Smokers and Non-smokers After Periodontal Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Cristiane Duque, PhD, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-26/103.243/2012
Record Dates: First submitted 2015-10-13; First posted 2015-10-20 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Periodontal Disease; Smoking
MeSH Terms: conditions — Periodontal Diseases; Smoking | interventions — Periodontal Index; Tooth Exfoliation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Periodontal treatment (Other): Both groups of patients (smokers and non-smokers) will receive periodontal treatment consisting of scaling and planning root, 4 times in the first month and after that once a month until complete one year. Patients will be clinically evaluated and microbiological collects will be made at baseline, 3 months, 6 months and 1 year after periodontal treatment.
  Interventions: Procedure: Periodontal treatment

INTERVENTIONS:
Procedure: Periodontal treatment — Periodontal treatment will consist of scaling and planning root, 4 times in the first month and after that once a month until complete one year. Patients will be clinically evaluated and microbiological collects were made at baseline, 3 months, 6 months and 1 year after periodontal treatment.
  Other Names: Scaling and planning root

SUMMARY:
Smoking has been considered the most important risk factor for periodontitis among all lifestyle factors. Fewer studies evaluated longitudinal clinical and microbiological status of smokers undergoing periodontal maintenance therapy and controversial results were found. This study will evaluate clinical conditions and prevalence of putative periodontopathogens and Candida spp. in smokers and non-smokers at baseline and after 3 and 6 months of nonsurgical periodontal therapy. Clinical parameters, including oral status assessed using Plaque Index (PI), Bleeding On Probe (BOP), Pocket Probing Depth (PPD), Gingival Recession (GR), Clinical Attachment Level (CAL) will be measured in smokers and non-smokers patients with chronic periodontitis. Samples of subgingival biofilm will be obtained from the periodontal pockets and furcation sites and submitted to phenol-chloroform DNA extraction and Polymerase Chain Reaction (PCR) analysis using specific primers for Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Prevotella intermedia, Campylobacter rectus, Candida albicans, Candida glabrata, Candida tropicalis and Candida dublinienses.

DETAILED DESCRIPTION:
Sixty patients (30 smokers (SM) and 30 non-smokers (NS) will be selected to participate of this study. All subjects will be recruited from the Department of Periodontology, School of Dentistry, Fluminense Federal University, Nova Friburgo, Rio de Janeiro State, Brazil. The study protocol was approved (protocol number: CAAE - 0070.0.258.000-10) by the Ethics Committee of the School of Medicine, Fluminense Federal University. Prior to participation, the purpose and procedures will be fully explained to all patients, who consequently gave written informed consent in accordance with the Helsinki Declaration. Medical and dental histories will be taken and patients will receive clinical evaluation at prescreening visits.

Clinical examination, microbiological collects and periodontal therapy Previous clinical examination, information about years of consumption of cigars and quantity of daily consumption will be recorded to select smokers and non- smokers subjects for the study. An experienced periodontist will perform clinical periodontal parameters in teeth for the protocol procedure. Each selected tooth selected will be measured for: Plaque Index (PI), Bleeding On Probe (BOP), Pocket Probing Depth (PPD), Gingival Recession (GR), Clinical Attachment Level (CAL) using a periodontal probe PCP15 (PCP-UNC15, Hu-Friedy, Chicago, IL), six sites (mesio-buccal, mediobuccal, disto-buccal, mesio-lingual, medio-lingual, disto-lingual) will be recorded. Sites with probing depth (PPD) > 5mm will be selected for microbiological analysis. After clinical measurements, the supragingival biofilm will be removed with sterile gauze. Gingival crevicular samples will be taken from 4 sites with the deepest PPD (>5mm) in each patient using a sterile paper point from the deepest pocket for 30s. Pooled biofilms from each site will be separated in two microtubes containing Tris -EDTA buffer (10 mM Tris-Hcl, 0.1 mM EDTA, pH 7.5) and were stored at -20°C. The samples will be analyzed microbiologically by Polymerase Chain Reaction - PCR. Periodontal treatment will be consisted of scaling and planning root, 4 times in first month and after that once a month until complete 1 year. Patients will be clinically evaluated and microbiological collects will be made at baseline, 3 months, 6 months and 1 year after periodontal treatment.

Microbiological evaluation - PCR assays DNA will be extracted and quantified in a spectrophotometer at 260 nm (Genesys 10UV, Rochester, NY, USA), in order to obtain a standard concentration of 100 ng/mL and stored at -20 °C for subsequent PCR reactions. Briefly, samples will be submitted to a lise solution (extraction buffer and proteinase K) and then purified using chloroform:isoamil-alcohol, followed by DNA precipitation with isopropanol and 70% ethanol. The DNA will be resuspended in TE buffer (10 mM Tris-HCl, 0.1 mM EDTA, pH 7.5, with 10 μg/mL RNAse). Microbial molecular identification will be carried out by PCR with specific primers for Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Prevotella intermedia, Campylobacter rectus, Candida albicans, Candida glabrata, Candida tropicalis and Candida dublinienses. PCR amplification will be performed with a GeneAmp PCR system 2400 (Perkin-Elmer - Applied Biosystems) for TGradient 96 (Biometra, Germany) under thermal conditions specific for each pair of primers. The PCR products will be separated by electrophoresis in 2% agarose gels and Tris-borate-EDTA running buffer (pH 8.0). The molecular mass ladder (100 bp DNA ladder, Gibco, Grand Island, NY, USA) will be included for running in the agarose gel. The DNA will be stained with 0.1µl of Sybr Safe/mL (Invitrogen, CA, USA) and visualized under UV illumination (Pharmacia LKB-MacroVue, San Gabriel, CA, USA). Photographs of the images will be taken (Image Mater - LISCAP, VDS, Pharmacia Biotech Piscataway, NJ, USA) and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* presence of periodontal disease in unirradicular teeth
* bleeding on probing in sites where probing depth was ≥5 mm in a minimum of two teeth in different arch;
* radiographic bone loss ranging from 30% to 50%.

Exclusion Criteria:

* patients with systemic diseases, diabetes; osteoporosis;
* pregnant lactating females;
* use of immune suppressive medication, phenytoin, cyclosporine, calcium channel blockers or any use of antibiotics or nonsteroidal anti-inflammatory drugs in the past 3 months;
* any medical conditions requiring immunotherapy or diagnosed as HIV+ or with AIDS, that could interfere with the periodontium status.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-01 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of periodontal status represented by means/standard deviations of the percentage of high scores of PI and BOP and levels (mm) of PPD, GR and CAL in smokers and non-smokers patients before and after periodontal treatment | Up to one year
  An experienced periodontist will perform clinical periodontal analysis and periodontal treatment. Six sites (mesio-buccal, mediobuccal, disto-buccal, mesio-lingual, medio-lingual, disto-lingual) of each selected tooth (at least six teeth) will be measured using standard scores for the following periodontal markers: Plaque Index (PI) and Bleeding On Probe (BOP) and determined the levels (mm) of Pocket Probing Depth (PPD), Gingival Recession (GR) and Clinical Attachment Level (CAL) using a periodontal probe PCP15 (PCP-UNC15, Hu-Friedy, Chicago, IL). Means/standard deviations will be calculated from the percentage of high scores of PI and BOP and levels (mm) of PPD, GR and CAL for each patient and after that for each group: smokers and non-smokers. All patients with periodontal disease (high scores of periodontal markers) will be submitted to periodontal treatment and clinically evaluated at baseline, 3 months, 6 months and 1 year after treatment.
Prevalence of periodontopathogens calculated in percentage of sites containing the species tested for PCR, comparing smokers and non-smokers | Up to one year
  Gingival crevicular samples will be taken from 4 sites with the deepest PPD (>5mm) in each patient. DNA from these samples will be extracted using phenol-chloroform method and quantified in a spectrophotometer at 260 nm and stored at -20 °C. Microbial molecular identification will be carried out by PCR with specific primers for Aggregatibacter actinomycetemcomitans, Porphyromonas gingivalis, Tannerella forsythia, Prevotella intermedia, Campylobacter rectus, Candida albicans, Candida glabrata, Candida tropicalis and Candida dublinienses. PCR amplification will be performed with a GeneAmp PCR system 2400 (Perkin-Elmer - Applied Biosystems) for TGradient 96 (Biometra, Germany) under thermal conditions specific for each pair of primers. The prevalence of periodontopathogens will be calculated in percentage of sites containing the species tested for PCR, comparing smokers and non-smokers at baseline, 3 months, 6 months and 1 year after periodontal treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Cristiane Duque, PhD, Principal Investigator — University of Sao Paulo; Gabriela AC Camargo, PhD, Study Director — Federal Fluminense University
Locations (1):
- Federal Fluminense University, Nova Friburgo, Rio de Janeiro, Brazil